CLINICAL TRIAL: NCT01289301
Title: Polyomavirus BK Nephropathy After Renal Transplantation: Randomized Clinical Trial to Demonstrate That Switching to mTOR Inhibitor is More Effective Than a Reduction of Immunosuppressive Therapy
Brief Title: Studying the Effect of Changing Immunosuppression in Case of Polyoma BK Virus Infection of the Renal Transplant
Acronym: BKVIRUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Clinical Research Center, Medizinische Hochschule
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Polyoma IFB 29
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2010-10

CONDITIONS: Disorder Related to Renal Transplantation; Immunosuppression Related Infectious Disease; Virus Diseases
Keywords: renal transplantation; polyoma BK virus infection; everolimus; calcineurin inhibitor; mTOR inhibitor
MeSH Terms: conditions — Virus Diseases | interventions — Sirolimus; Everolimus; Cyclosporine; Tacrolimus; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mTOR-receiving arm (Experimental): switching from calcineurin-inhibitor-based immunosuppression to mTOR-based immunosuppression
  Interventions: Drug: mTOR inhibitor (everolimus)
- calcineurin-inhibitor keeping arm (Active Comparator): continuing calcineurin-inhibitor based immunosuppression
  Interventions: Drug: cyclosporine or tacrolimus

INTERVENTIONS:
Drug: mTOR inhibitor (everolimus) — calcineurin-inhibitor based immunosuppression will be switched to immunosuppression based on m-TOR inhibitor (everolimus trough level 3-7ng/mL)
  Other Names: switch immunosuppression to everolimus
  Arms: mTOR-receiving arm
Drug: cyclosporine or tacrolimus — calcineurin inhibitor (cyclosporine or tacrolimus) will be continued (trough level 60-90ng/mL resp 3-7ng/mL)
  Other Names: keeping immunosuppression with calcineurin inhibitor; cyclosporine; tacrolimus
  Arms: calcineurin-inhibitor keeping arm

SUMMARY:
Polyomavirus BK nephropathy is a serious complication after renal transplantation leading to graft loss in 40% of cases. Since no virustatic drug exists, the investigators want to study the best way to manage viral invasion by changing the immunosuppressive treatment comparing two treatment schemes. The investigators hypothesis is that switching to an mTOR-based scheme is superior to a general decrease of a calcineurin inhibitor (CNI)-based scheme. The study will be performed as a prospective, randomized, parallel group comparison.

DETAILED DESCRIPTION:
The study group (n=62) will be switched from CNI to everolimus while the control group (n=62) will get a general reduction of the CNI-based immunosuppression. Follow-up and duration of intervention per patient will be 24 months, duration of the trial 72 months including 4 years of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* preceding renal transplantation
* functioning graft with a permanent creatinine clearance of more than 25mL/min
* biopsy-confirmed polyoma BK virus nephropathy
* age over 18 years old

Exclusion Criteria:

* allergy or non-tolerance of the study medication everolimus
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
death or graft loss | 2 years of observation
  after experimental intervention (switch to mTOR inhibitor in group 1) and control intervention (general reduction of immunosuppression) observation of graft function

SECONDARY OUTCOMES:
decrease of polyomavirus serum PCR | 2 years
  regular measurement of polyomavirus serum PCR (every 4 weeks to 3 months)
decrease of creatinine | 2 years observation
  regular measurment of graft function (every 4 weeks to 3 months)
progression of chronic changes in renal histology | renal biopsy 3 months after intervention
  renal rebiopsy and comparison of chronic changes in renal biopsy with the diagnostic renal biopsy
number of rejections following intervention | 2 years after intervention
  biopsy-verified rejections (graft biopsies on indication) may be a consequence of changement of immunosuppression and a side effect of it, rejections will be counted
increase of BKV-specific T-cells | 2 years observation
  increase of BKV-specific T-cells are a sign of overcoming viral infection and will be counted regularly (every 3 to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Anke Schwarz, Prof. Dr., Principal Investigator — Hannover Medical School, Nephrology; Hermann Haller, Prof. Dr., Principal Investigator — Hannover Medical School, Nephrology; Silvia Linnenweber, Dr., Study Chair — Hannover Medical School, Nephrology; Armin Koch, Prof. Dr., Study Director — Hannover Medical School, Biometry; Albert Heim, PD Dr., Study Director — Hannover Medical School, Virology; Verena Broecker, Dr., Study Chair — Hannover Medical School, Pathology
Locations (4):
- Germany (4):
  - University Hospital Freiburg, Transplant Outpatient Clinic, Freiburg im Breisgau, Baden-Wurttemberg
  - University of Erlangen/ Nürnberg, Transplant Outpatient Clinic, Erlangen, Bavaria
  - Hannover Medical School, Transplant Outpatient Clinic, Hanover, Lower Saxony
  - University of Essen, Transplant Outpatient Clinic, Essen, Ruhrgebiet